CLINICAL TRIAL: NCT04782544
Title: Assessing Whether Buttermilk Powder Improves Disease Activity in Pediatric IBD
Brief Title: Ganglioside and IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Orange County (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 200109
Record Dates: First submitted 2021-02-23; First posted 2021-03-04 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2022-07

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Active Comparator): 5 grams of buttermilk powder daily for 10 weeks, oral.
  Interventions: Other: Buttermilk Powder
- Placebo (Placebo Comparator): 5 grams of milk powder (10% buttermilk powder, 90% anhydrous milk fat) daily for 10 weeks, oral.
  Interventions: Other: Anhydrous Milk Fat

INTERVENTIONS:
Other: Buttermilk Powder — Treatment with 5.0 g of buttermilk powder daily for 10 weeks.
  Arms: Treatment
Other: Anhydrous Milk Fat — Treatment with 5.0 g of milk powder (90% anhydrous milk fat, 10% buttermilk powder) daily for 10 weeks.
  Arms: Placebo

SUMMARY:
Context. Inflammatory bowel disease (IBD) is a chronic and debilitating disorder. Novel treatment strategies aimed to resolve intestinal inflammation and induce disease remission are necessary. Dietary gangliosides are safe for consumption, bioavailable, and have shown clinical benefit in patients with inflammatory intestinal disease.

Objectives. The primary objective is this study is to determine the efficacy of dietary ganglioside in improving disease activity indices in pediatric patients with IBD. Secondary objectives include demonstrating the effectiveness of dietary ganglioside for improving quality of life, improving intestinal integrity, and reducing inflammation.

Study Design. Intervention: controlled trial (pilot). Participants. Inclusion criteria: aged 9-21 years, diagnosis of ulcerative colitis (UC) or ileal or colonic Crohn Disease (CD), active disease. Exclusion criteria: pregnancy, inadequate liver or renal function, active infectious disease, previous bowel resection, disease remission, drug/alcohol abuse, other serious medical conditions, indeterminate colitis.

Study Intervention. Patients with IBD (n=48) will be allocated to consume ganglioside treatment or placebo daily for 10 weeks. Treatment group will consume five grams of buttermilk powder daily or anhydrous milk fat.

Outcome Measures. The primary outcome is the disease activity index: pediatric Crohn's Disease Activity Index (pCDAI) or pediatric Ulcerative Colitis Activity Index (pUCAI). Secondary outcomes include: quality of life (IMPACT-III questionnaire), intestinal permeability (lactulose/mannitol urinary assay), C-reactive protein (CRP; blood exam), calprotectin (fecal exam).

Expected Outcomes. Relative to the placebo group, the treatment group will have improved disease activity indices, quality of life, and intestinal integrity over the 10-week study period. The treatment group will also show reduction in inflammation and calprotectin relative to the placebo group.

ELIGIBILITY:
Inclusion Criteria:

1. Participants age 9-21 years
2. Mild-moderate IBD defined by ImproveCareNow (ICN) Physician Global Assessment (PGA); OR severe IBD defined by ICN PGA if stable for at least 120 days
3. Ileal, ileocolonic, colonic location of disease

Exclusion Criteria:

1. Pregnancy
2. Previous bowel resection
3. Non-ileocolonic location of disease
4. Inadequate liver or renal function
5. On prescription medication for active infectious disease
6. Drug/alcohol abuse
7. Other serious medical conditions

Ages: 9 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2024-03-24 (Actual)

PRIMARY OUTCOMES:
Disease activity index | Day 0
  Pediatric 1) Crohn Disease or 2) Ulcerative Colitis disease activity index
Disease activity index | Day 70
  Pediatric 1) Crohn Disease or 2) Ulcerative Colitis disease activity index

SECONDARY OUTCOMES:
ImproveCareNow Physician Global Assessment | Day 0
  A disease activity index
ImproveCareNow Physician Global Assessment | Day 70
  A disease activity index
IMPACT-III questionnaire | Day 0
  quality of life scales (0 = lowest, 100 = highest): well-being, emotional functioning, social functioning, body image
IMPACT-III questionnaire | Day 70
  quality of life scales (0 = lowest, 100 = highest): well-being, emotional functioning, social functioning, body image
Intestinal integrity | Day 0
  Intestinal permeability (lactulose/mannitol) challenge
Intestinal integrity | Day 70
  Intestinal permeability (lactulose/mannitol) challenge
Calprotectin | Day 0
  Stool test
Calprotectin | Day 70
  Stool test
C-reactive protein | Day 0
  Blood test
C-reactive protein | Day 70
  Blood test

OTHER OUTCOMES:
Hemoglobin, study start | Day 0
  g/L, from metabolic panel
Hemoglobin, study end | Day 70
  g/L, from metabolic panel
Platelets, study start | Day 0
  #, from metabolic panel
Platelets, study end | Day 70
  #, from metabolic panel
White blood cells, study start | Day 0
  #, from metabolic panel
White blood cells, study end | Day 70
  #, from metabolic panel
Albumin, study start | Day 0
  g/L, from metabolic panel
Albumin, study end | Day 70
  g/L, from metabolic panel
Hematocrit, study start | Day 0
  proportion, from metabolic panel
Hematocrit, study end | Day 70
  proportion, from metabolic panel

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Orange County, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No